CLINICAL TRIAL: NCT05564221
Title: A Randomized, Double-Blind, Placebo/Active Controlled, Multiple Ascending Dose, Phase 1b Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics Following Subcutaneous Injections of YH35324 in Atopic Healthy Subjects or Subjects With Allergic Diseases
Brief Title: A Multiple Ascending Dose, Phase 1b Study of YH35324 in Atopic Healthy Subjects or Subjects With Allergic Diseases
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yuhan Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: YH35324-102
Record Dates: First submitted 2022-09-19; First posted 2022-10-03 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2024-12

CONDITIONS: Atopic Healthy Subjects; Adult Subjects With Allergic Diseases
Keywords: GI-301; YH35324; Allergic disease
MeSH Terms: interventions — Omalizumab; Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: As the YH35324 group and placebo group will be double-blinded, YH35324 and placebo will have the same appearance and packaging. Therefore, the double-blind will apply to the subjects, investigators, study coordinators, and study personnel including study pharmacists.
  The active control omalizumab has a different appearance and packaging from YH35324 and placebo, and will be administered in an open-label manner.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- YH35324 (Experimental): There will be 5 dose groups of YH35324, escalating from low to high doses in a stepwise manner: Cohort 1(A mg/kg) → Cohort 2(B mg/kg) → Cohorts 3(C mg/kg) and 4(C mg/kg) → Cohort 5(C mg/kg) YH35324 and placebo will be administered in a double-blinded manner.
  Interventions: Drug: YH35324
- Placebo (Placebo Comparator): There will be 5 dose groups of YH35324, escalating from low to high doses in a stepwise manner: Cohort 1(A mg/kg) → Cohort 2(B mg/kg) → Cohorts 3(C mg/kg) and 4(C mg/kg) → Cohort 5(C mg/kg) YH35324 and placebo will be administered in a double-blinded manner.
  Interventions: Drug: Placebo
- Omalizumab (Active Comparator): For Cohort 3, omalizumab 300 mg will be administered in an open-label manner.
  Interventions: Drug: Omalizumab

INTERVENTIONS:
Drug: YH35324 — Subcutaneous injection of YH35324
  Arms: YH35324
Drug: Placebo — Subcutaneous injection of None of active ingredient
  Arms: Placebo
Drug: Omalizumab — Subcutaneous injection of Omalizumab
  Other Names: Xolair® prefilled syringe 150 for injection
  Arms: Omalizumab

SUMMARY:
This study aims to evaluate the safety, tolerability, pharmacokinetic (PK) and pharmacodynamic (PD) profiles following multiple subcutaneous injections of YH35324 in healthy subjects or subjects with allergic diseases, who have atopy.

DETAILED DESCRIPTION:
YH35324 is a drug under development as a novel therapeutic agent for various IgE-mediated allergic diseases. Since YH35324 has a high binding affinity to human IgE, it prevents serum IgE from binding to receptors on mast cells and basophil, thereby inhibiting histamine release caused by degranulation when exposed to allergens. This study aims to evaluate the safety, tolerability, pharmacokinetic (PK) and pharmacodynamic (PD) profiles following multiple subcutaneous injections of YH35324 in healthy subjects or subjects with allergic diseases, who have atopy.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adults aged ≥ 19 to ≤ 55 years(Cohort 5, Mald or female adults ≥ 19)
* Serum total IgE level ≥ 30 IU/mL or 30 to 700 IU/mL or >700IU/mL(Not Applicable for Cohort 5)
* Meeting the following cohort-specific disease severity criteria [Cohorts 1-4]: Healthy subjects without any pathological symptoms or findings from medical examination, or subjects with a history of mild allergic diseases (allergic rhinitis, atopic dermatitis, food allergy, urticaria, or allergic asthma) [Cohort 5]: Subject who have been diagnosed with moderate to severe atopic dermatitis

Exclusion Criteria:

* History of malignancy
* Positive drug screen result
* transaminase (AST) or alanine transaminase (ALT) level > 2 X the upper limit of normal
* Estimated glomerular filtration rate (eGFR) < 60 mL/min/1.73 m2 using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula
* Allergy immunotherapy initiated or changed within 6 months prior to randomization(For Cohort 5, within 12 months prior to randomization)
* History of participation in another clinical trial within 6 months prior to randomization

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-11-28 (Actual); Study Completion 2024-11-28 (Actual)

PRIMARY OUTCOMES:
Occurrence and severity of adverse events (AEs) | Occurrence and severity of adverse events will be observed for 141 days after administration in Cohorts 1 to 5
  To evaluate the safety and tolerability following multiple administrations of YH35324

SECONDARY OUTCOMES:
Area Under the Serum Concentration-Time Curve from Zero to the Time of the Last Quantitative Concentration (AUClast) | Serum concentrations of YH35324 will be observed for 141 days after administrationin in Cohorts 1 to 4
  To evaluate the PK profile of YH35324
Area Under the Serum Concentration-Time Curve from Zero to Infinity (AUCinf) | Serum concentrations of YH35324 will be observed for 141 days after administration in Cohorts 1 to 4
  To evaluate the PK profile of YH35324
Maximum Serum Concentration(Cmax) | Serum concentrations of YH35324 will be observed for 141 days after administration in Cohorts 1 to 4
  To evaluate the PK profile of YH35324
Time to Maximum Serum Concentration (Tmax) | Serum concentrations of YH35324 will be observed for 141 days after administration in Cohorts 1 to 4
  To evaluate the PK profile of YH35324
Terminal Elimination Rate Constant, Apparent Terminal Elimination Half-life (t1/2) | Serum concentrations of YH35324 will be observed for 141 days after administration in Cohorts 1 to 4
  To evaluate the PK profile of YH35324
Apparent Serum Clearance (CL/F) | Serum concentrations of YH35324 will be observed for 141 days after administration in Cohorts 1 to 4
  To evaluate the PK profile of YH35324
Apparent Volume of Distribution (Vz/F) | Serum concentrations of YH35324 will be observed for 141 days after administration in Cohorts 1 to 4
  To evaluate the PK profile of YH35324
Area Under the Serum Concentration-Time Curve during dosing interval at steady-state (AUCtau) | Serum concentrations of YH35324 will be observed for 141 days after administration in Cohorts 1 to 4
  To evaluate the PK profile of YH35324
Maximum Serum Concentration at steady-state (Cmax,ss) | Serum concentrations of YH35324 will be observed for 141 days after administration in Cohorts 1 to 4
  To evaluate the PK profile of YH35324
Time to Maximum Serum Concentration at steady-state (Tmax,ss) | Serum concentrations of YH35324 will be observed for 141 days after administration in Cohorts 1 to 4
  To evaluate the PK profile of YH35324
Accumulation ratio (Rac) | Serum concentrations of YH35324 will be observed for 141 days after administration in Cohorts 1 to 4
  To evaluate the PK profile of YH35324
Change in serum free IgE level | Change in serum Free IgE will be observed for 141 days after administration in Cohorts 1 to 5
  To evaluate the PD profile on serum IgE following multiple administrations of YH35324
Change in serum total IgE level | Change in serum Total IgE will be observed for 141 days after administration in Cohorts 1 to 4
  To evaluate the PD profile on serum IgE following multiple administrations of YH35324
Serum concentrations of YH35324 | Serum concentrations of YH35324 will be observed for 99 days after administration in Cohorts 5
  To evaluate the PK profile of YH35324
Change in Eczema Area and Severity Index (EASI) | Change in Eczema Area and Severity Index (EASI) will be observed for 141 days after administration in Cohorts 5
  To explore the clinical efficacy following multiple administrations of YH35324
Change in Validated Investigator Global Assessment (vIGA-AD) | Change in Validated Investigator Global Assessment (vIGA-AD) will be observed for 141 days after administration in Cohorts 5
  To explore the clinical efficacy following multiple administrations of YH35324
Change in SCORing Atopic Dermatitis (SCORAD) | Change in SCORing Atopic Dermatitis (SCORAD) will be observed for 141 days after administration in Cohorts 5
  To explore the clinical efficacy following multiple administrations of YH35324
Change in Pruritus-Numerical Rating Scale (NRS) | Change in Pruritus-Numerical Rating Scale (NRS) will be observed for 141 days after administration in Cohorts 5
  To explore the clinical efficacy following multiple administrations of YH35324
Change in body surface area (BSA) of atopic dermatitis involvement | Change in body surface area (BSA) of atopic dermatitis involvement will be observed for 141 days after administration in Cohorts 5
  To explore the clinical efficacy following multiple administrations of YH35324
Number of days of rescue treatment (TCS or TCI) used | Number of days of rescue treatment (TCS or TCI) used will be observed for 141 days after administration in Cohorts 5
  To explore the clinical efficacy following multiple administrations of YH35324

OTHER OUTCOMES:
Changes in FcεRI expression on basophil surface | Changes in FcεRI expression will be observed for 141days after administrationin in Cohorts 1 to 4
  To explore the PD profile on serum basophil following multiple administrations of YH35324
Changes in allergen-induced skin prick wheal response | Changes in allergen-induced skin prick wheal response will be observed for 113 days in Cohorts 1 to 5
  To explore inhibition on allergens (allergy antigens) following multiple administrations of YH35324
Changes in serum allergen specific IgE level | Changes in allergen-induced serum allergen specific IgE level will be observed for 141 days after administration in Cohorts 1 to 5
  To explore inhibition on allergens (allergy antigens) following multiple administrations of YH35324
Incidence of serum anti-YH35324 antibodies | Incidence of serum Anti-YH35324 antibodies will be observed for 141 Days after administration in Cohorts 1 to 5
  To explore the immunogenicity following multiple administrations of YH35324
Changes in serum Thymus and Activation-Regulated Chemokine (TARC, CCL17) and Macrophage-Derived Chemokine (MDC, CCL22) | Changes in serum Thymus and Activation-Regulated Chemokine and Macrophage-Derived Chemokine will be observed for 141 Days after administration in Cohorts 5
  To explore the PD following multiple administrations of YH35324
Changes in serum cytokines (IL-4, IL-5, IL-10, IL-18, IL-22, IL-13, IL-31, IL-33, and IFN-γ) levels | Changes in serum cytokines levels will be observed for 141 Days after administration in Cohorts 5
  To explore the PD following multiple administrations of YH35324

CONTACTS AND LOCATIONS:
Overall Officials: Hae-Sim Park, Study Chair — Ajou University School of Medicine
Locations (9):
- South Korea (9):
  - Soonchunhyang University Bucheon Hospital, Bucheon-si, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Ajou University Hospital, Suwon, Gyeonggi-do
  - Nowon Eulji Medical Center, Seoul
  - Korea University Anam Hospital, Seoul
  - Severance Hospital, Seoul
  - Konkuk University Medical Center, Seoul
  - Asan Medical Center, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (including data dictionaries) that underline the results reported in study-related publications will be made available during the period beginning 1 year and ending 5 years after all trial primary and secondary endpoints were assessed. Only requests from researchers who provide a methodologically sound proposal will be reviewed and approved by the sponsor. The analysis type should be in accordance with aims in the proposal approved by the sponsor. Proposals should be directed to yhcho@yuhan.co.kr.
  A summary of the study results will be posted in the publicly accessible database (i.e. clinicaltrials.gov) no later than 1 year after the study's primary completion date.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Beginning 1 year and ending 5 years after all trial endpoints were assessed
Access Criteria: Only requests from researchers who provide a methodologically sound proposal will be reviewed and approved by the sponsor. The analysis type should be in accordance with aims in the proposal approved by the sponsor. Proposals should be directed to yhcho@yuhan.co.kr